CLINICAL TRIAL: NCT02358421
Title: High Response Predictive Parameters After Controlled Ovarian Stimulation in Women Undergoing Assisted Reproductive Techniques
Brief Title: Prediction of High Ovarian Response After Assisted Reproductive Techniques
Acronym: HighART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: Highresponse_ART
Record Dates: First submitted 2014-03-21; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: PCOS; OHSS
Keywords: Rotterdam's diagnostic criteria of PCOS; Risk of OHSS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Initial cohort: Patients at risk of developing OHSS according to the inclusion criteria

SUMMARY:
Polycystic ovarian syndrome (PCOS) patients have an increased risk of ovarian hyperstimulation syndrome (OHSS) after assisted reproduction techniques (ART). In addition, these women have a high risk of develop further metabolic disorders. Rotterdam criteria defined by the European Society of Human Reproduction and Endocrinology (ESHRE) are used for the diagnosis of PCOS.

The aim of this study is both to determine the prevalence of PCOS in infertile patients who require ART in our Center and to evaluate the usefulness of each specific diagnosis criterium within Rotterdam criteria of PCOS as predictor of risk of OHSS. It also seeks to establish a cohort of patients identified according to specific Rotterdam criteria of PCOS to assess the incidence of long term complications.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women. It affects 10 % of patients who undergo assisted reproductive techniques (ART). Rotterdam criteria defined by the European Society of Human Reproduction and Endocrinology (ESHRE) are used for the diagnosis of PCOS. According to such criteria, PCOS affects 5-10% of women of reproductive age.

Patients with PCOS according to the Rotterdam criteria, as well as those with polycystic ovaries by ultrasound, have a high risk of an exaggerated response to ovulation induction therapy. Complications of the ovarian hyperstimulation syndrome (OHSS) include hemoconcentration, thromboembolic disorders, electrolyte disorders, ascites, hydrothorax, ovarian torsion, respiratory failure, liver failure, kidney failure or even death.

There is a lack of reliable markers that indicate risk of OHSS. It is also unknown whether any specific criteria proposed in the Rotterdam consensus is more important than another or independently influence on the results of the ARTs.

The aim of this study is both to determine the prevalence of PCOS in infertile patients who require ART in our Center and to evaluate the usefulness of each specific diagnosis criteria of PCOS as predictor of risk of OHSS. It also seeks to establish a cohort of patients identified according to specific Rotterdam criteria of PCOS to assess the incidence of long term complications.

ELIGIBILITY:
Inclusion criteria:

Patients with primary infertility undergoing ovarian stimulation for IVF/ICSI plus one of the following criteria:

1. Ovulation dysfunction.
2. Androgen excess: clinical and/or biochemical.
3. Polycystic ovary by transvaginal ultrasound in early follicular phase.
4. AMH>35 pmol/l
5. FSH/LH<1
6. P4 levels on the day of menstrual cycle <10ng/ml and cycle duration <26 days
7. Patients who undergo a second cycle after a previous one in which they were considered high responders (the cycle was canceled due to high risk of OHSS or the patient underwent coasting)

Exclusion Criteria:

1. Age <18 or >39 years
2. FSH >10
3. Uterine fibroids requiring surgery
4. Diagnosis of hyperprolactinemia , hypothyroidism, congenital adrenal hyperplasia, Cushing's syndrome, ovarian tumors, adrenal tumors or hypogonadotropic hypogonadism
5. Intake of oral contraceptives three months prior to the completion of IVF
6. Diagnosis of endometriosis (by ultrasound or surgical findings)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with primary infertility at risk of developing ovarian hyperstimulation syndrome during controlled ovarian hyperstimulation. This population was defined according to the presence of at least one Rotterdam criterion or the presence of an abnromal luteal phase, invesion of the FSH/LH ratio or an increased AMH level (see inclusion and exclusion criteria below)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, negative and positive predictive values of each inclusion criteria (independently and combined) to predict OHSS and high ovarian response after ART | 18 months

SECONDARY OUTCOMES:
Prevalence of metabolic syndrome in the cohort of included patients | After COH for ART
  18 months
Incidence of metabolic syndrome in patients with at least one criterion of PCOS | 15 years in average
Incidence of cardiiovascular events in patients with at least one criterion of PCOS | 15 years in average

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Montañana-Ramirez, MD, PhD, Principal Investigator — Instituto de Investigaciones Sanitarias La Fe
Locations (1):
- La Fe University Hospital, Valencia, Valencia, Spain